CLINICAL TRIAL: NCT03439423
Title: Controllo Dopo Trattamento Endovascolare di Aneurismi Aortici Mediante Risonanza Magnetica Senza Mezzo di Contrasto ed Ecografia Con Color-doppler: Accuratezza Diagnostica, Analisi Costo-efficacia e Impatto Sul Management Del Paziente
Brief Title: Control Post Endovascular Treatment of Aortic Aneurisms Through Magnetic Resonance and Ultrasound (SAFEVAR)
Status: Completed | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Francesco Sardanelli, Head of Radiology Department, IRCCS Policlinico S. Donato
Other Study IDs: SAFEVAR_v02
Record Dates: First submitted 2018-02-02; First posted 2018-02-20 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Abdominal Aortic Aneurism
MeSH Terms: interventions — Contrast Media; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who underwent EVAR
  Interventions: Radiation: CT with contrast agent; Diagnostic Test: MR without contrast agent; Diagnostic Test: Color-Doppler Ultrasound; Other: Questionnaire

INTERVENTIONS:
Radiation: CT with contrast agent
Diagnostic Test: MR without contrast agent — on 1.5-T unit, with the following sequences:
  * steady-state free-precession (true-FISP)
  * half-Fourier single shot spin-echo (HASTE)
Diagnostic Test: Color-Doppler Ultrasound
Other: Questionnaire — regarding their perception of examinations

SUMMARY:
The aims of this study are to verify non-inferiority of magnetic resonance (MR) without contrast agent associated to color-Doppler ultrasound for the diagnosis of endoleaks after endovascular aortic repair (EVAR), to evaluate both the economical and biological cost-effectiveness of such diagnostic algorithm as an alternative to computed tomography (CT) with contrast agent, and to analyze its impact on both patients work-flow and infrastructure logistics

DETAILED DESCRIPTION:
In this prospective observational study, 250 patients who underwent EVAR will be studied. They will be enrolled after referral for a CT with contrast agent at IRCCS Policlinico San Donato or at ASST Santi Paolo e Carlo. Those with absolute contraindications to RM will be excluded.

All enrolled subjects will undergo MR with contrast agent and color-Doppler ultrasound after CT. Before and after each examination, they will be submitted a questionnaire to evaluate their perception towards the former, and both costs and exposure deriving from such examinations will be evaluated along with patients' responses. Moreover, both CT and MR along with color-Doppler ultrasound will be analyzed with regards to human resources management, operational management, patients' clinical workflow and organization.

All CT examinations will be independently evaluated by two radiologists with 4- and 8-year expertise in thoracic or abdominal CT. Results obtained from CT examinations will be used as a reference standard using the "worst case scenario" method: if either reader reported endoleak, the CT will be considered positive. The more experienced reader will anonymously and randomly repeat CT evaluation after 1 month.

For CMR examinations, a 15-minute protocol will be used on a 1.5-T device. The following sequences will be performed:

* steady state free-precession (true-FISP)
* half-Fourier single shot spin-echo (HASTE) All examinations will be independently and blindly evaluated by the same two radiologists as CT examinations, and they will be considered positive if areas (even smaller than 5 mm) of alterate signal in comparison to surrounding muscle in the same slice are present inside the aneurismatic sac. The more experienced reader will anonymously and randomly repeat CT evaluation after 1 month.

Color-Doppler ultrasound will be performed with a 1-5 MHz probe, by a radiologist with 7-year expertise in aortic ultrasound, blinded to MR and CT results. Ultrasound images will be evaluated both directly and through spectral flow study.

The sample size was calculated assuming an alpha error of 5%, 90% power and 10% endoleak prevalence. In order to prove a negative predictive value of MR without contrast agent and color-Doppler ultrasound not inferior to 90%, 250 patients should be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18
* informed written consent
* with either thoracic or abdominal aortic endoprosthesis

Exclusion Criteria:

* lack of informed written consent
* patients with absolute contraindications to magnetic resonance imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent endovascular aortic repair
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2016-03-09 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-09-12 (Actual)

PRIMARY OUTCOMES:
Sensitivity and negative predictive value | 2 year
  CT exams with contrast agent will be interpreted by 2 independent and blinded radiologists. The results of enhanced CT will be used as reference standard basing to "worst case scenario" method, i.e. it will be considered positive when one or both readers will report the presence of endoleak. Moreover, in the same way, the most expert reader will repeat the reading after 1 month compared to the first reading. Enhanced 1.5-T MRI will be conducted using true-FISP and HASTE sequences.
  The same 2 readers will evaluate the exams comparing to the previous CT exams. Images will be considered positive for the presence of endoleak if inside the aneurysmal sac excluded there will be an area of altered signal compared to adjacent muscles displayed in the same layers. The most experienced reader will repeat the exam reading 1 month later.
  The 1,5 MHz Color-Doppler ultrasound will be performed by a radiologist with 7 y of experience in vascular ultrasound of the aorta, blinded to the enhanced CT.

SECONDARY OUTCOMES:
Efficacy of the two diagnostic approaches | 2 year
  A systematic review of the literature will be performed and the data will be used to compare the efficacy of the two diagnostic approaches.
Patient's perception | 2 year
  To evaluate and compare the patient's perception of the examination performed (both MR and CT-free MCD and CT), we will use a EuroQoL5 questionnaire. Patients will be asked to complete the questionnaire before and after each survey. Regarding the economic costs, we will compare the main medical costs (equipment, drugs, used devices, personnel, etc.) to complete the two different diagnostic strategies compared.
Economic costs | 2 year
  Regarding the economic costs, we will compare the main medical costs (equipment, drugs, used devices, personnel, etc.) to complete the two different diagnostic strategies compared.
Patient management | 2 year
  To investigate how the introduction of new technologies in the health field questions the traditional organizational dynamics, two treatments will be examined and compared in terms of human resources, operational management of the treatment process, clinical pathway of the patient and organizational structure.
Involvement of professionals | 2 year
  All the professionals involved in the new diagnostic strategy will be interviewed to identify the organizational strengths and weaknesses related to the new diagnostic strategy in order to allow ad-hoc interventions to improve the process.
Patient acceptance and satisfaction | 2 year
  Regarding the level of patient acceptance and satisfaction, a questionnaire will be proposed and, the results will provide important information to identify the strengths and weaknesses of the treatment and to refine the procedure in order to maximize patient satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided